CLINICAL TRIAL: NCT02738229
Title: Should We Use Oral Valacyclovir in Acute Herpetic Gingivostomatitis in Children? A Randomized Controlled Trial
Brief Title: Should We Use Oral Valacyclovir in Acute Herpetic Gingivostomatitis in Children?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Association of Emergency Physicians (Industry)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, MSc, FRCPC, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Valtrex for HGS
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Herpetic Gingivostomatitis
MeSH Terms: conditions — Stomatitis, Herpetic | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valacyclovir (Experimental): Valacyclovir will be given twice a day with following doses according to weight:
  10 to 13,9 kg : Valacyclovir 250 mg PO twice per day 14 to 19,9 kg : Valacyclovir 375 mg PO twice per day 20 to 28 kg : Valacyclovir 500 mg PO twice per day
  Interventions: Drug: Valacyclovir
- control (Placebo Comparator): placebo pill
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Valacyclovir
  Arms: Valacyclovir
Drug: placebo
  Arms: control

SUMMARY:
Primary herpetic gingivostomatitis is a frequent problem in pediatrics. Complications of this are dehydration, pain and hospitalisation. The objective of this randomized controlled trial is to assess the clinical efficacy of oral Valacyclovir to decrease the duration of symptoms associated with acute herpes gingivostomatitis in children. This study will involve 80 children aged 1 to 8 years old to receive weight adjusted doses of valacyclovir for 7 days. The primary outcome measure will be the duration (in days) of feeding and/or drinking difficulties.

ELIGIBILITY:
Inclusion criteria are :

* Children from 10 to 28 Kg of weight. The inclusion of participants is based on weight for practical/feasibility reasons because the study medication will be provided in tablet format. The lower limit of 10 kg is to limit to three strata of weight and limit costs engendered by the preparation of medication.
* Clinical diagnosis of herpetic gingivostomatitis according to the treating physician. This is described by the presence of:

  * Fever (>38.5° rectal, >38° oral) AND
  * Vesicular or ulcerative lesions located in the anterior of the mouth
  * Associated or not with perioral vesicular lesions Visiting the emergency department within the first 96 hours of the disease begin.

Exclusion criteria are :

* Duration of fever > 4 days
* Hospitalised patients
* Immunocompromised patients
* Patients with known hypersensitivity to Valacyclovir
* Patients with renal failure
* Children with complete incapacity of oral treatment intake
* Unable to be contacted for phone follow-up

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-07; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Duration of feeding and/or drinking difficulties | 2 weeks
  This will be defined by the number of days until the participants return to normal feeding and eating according to the parents.

SECONDARY OUTCOMES:
duration of fever | 2 weeks
duration of pain | 2 weeks
duration of oral lesions | 2 weeks
global parent satisfaction | 2 weeks
  Likert scale on how satisfied the parents are with the medication. This will be measured during a follow-up survey at 7 and 14 days following randomisation
duration of school or work absence | 2 weeks
utilisation of medical resources | 2 weeks
  hospitalisation for intra venous hydration, visit to a physician, use of analgesics or other medication. This will be measured during a follow-up survey at 7 and 14 days following randomisation
adverse side effects | 2 weks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided